CLINICAL TRIAL: NCT06436053
Title: Acute Response to Left Bundle Branch Area Pacing With SyncAV
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10516
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- LBBAP with SyncAV
  Interventions: Device: LBBAP with SyncAV

INTERVENTIONS:
Device: LBBAP with SyncAV — Acute changes in surface ECG QRS duration resulting from left bundle branch area pacing using various pacing configurations will be evaluated.

SUMMARY:
This clinical investigation is a prospective, single-arm, post-market, non-randomized, single-center study designed to evaluate the effectiveness of the SyncAV CRT dynamic atrioventricular (AV) delay feature when used with left bundle branch area pacing (LBBAP).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age and willing to comply with the study requirements
2. Patients with approved indication for dual-chamber pacing or cardiac resynchronization therapy and scheduled to be implanted with an Abbott pacing system
3. Patient has documented left bundle branch block (LBBB) or intraventricular conduction delay (IVCD)
4. Patient has an intrinsic QRS duration ≥ 130 ms
5. Patient has intact AV conduction with PR interval ≤ 250 ms

Exclusion Criteria:

1. Patient has a resting ventricular rate > 100 bpm
2. Patient has AV Block (2nd or 3rd degree)
3. Patient has documented persistent atrial tachycardia or atrial fibrillation
4. Patient has had a recent myocardial infarction, ablation, electrolyte imbalance, or any condition within the last 90 days that would contraindicate for pacing device programming changes in the opinion of the investigator
5. Patient is currently participating in another clinical investigation
6. Patient is pregnant or nursing
7. Patient has other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
8. Patient does not have legal authority
9. Patient is unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with approved indication for dual-chamber pacing or cardiac resynchronization therapy, with documented left bundle branch block or intraventricular conduction delay, long QRS duration, and intact AV conduction will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
QRS duration | During the intervention/procedure/surgery
  Acute change in surface ECG QRS duration resulting from left bundle branch area pacing with optimized SyncAV, relative to intrinsic atrioventricular conduction.

SECONDARY OUTCOMES:
LV hemodynamics | During the intervention/procedure/surgery
  Acute change in left ventricular hemodynamics (i.e., maximum rise in pressure) resulting from left bundle branch area pacing with optimized SyncAV, relative to intrinsic atrioventricular conduction.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No